CLINICAL TRIAL: NCT01480960
Title: Effects of a Whole Body Vibration Training on the Exercise Performance in Patients After Lung Transplantation
Brief Title: Effects of a Whole Body Vibration Training in Patients After Lung Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Dr. med. Klaus Kenn, Head physician, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTX2011
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Patients Following Lung Transplantation (Single and Double)
Keywords: lung transplantation; whole body vibration; exercise training; pulmonary rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole body vibration training (Active Comparator): Whole body vibration training in addition to pulmonary rehabilitation
  Interventions: Other: Pulmonary rehabilitation + whole body vibration training
- No whole body vibration training (No Intervention): Pulmonary rehabilitation without whole body vibration training

INTERVENTIONS:
Other: Pulmonary rehabilitation + whole body vibration training — standard inpatient rehabilitation program including endurance and strength plus squats on a vibration plate for 4x2 minutes, 3 times per week
  Other Names: Galileo training
  Arms: Whole body vibration training

SUMMARY:
Pulmonary rehabilitation has been established as an evidence-based and recommended therapy in patients following lung transplantation. Exercise training has been shown to be a cornerstone of an inpatient rehabilitation program to reduce muscle dysfunction and improve exercise performance. In our study we will investigate the benefit of a whole body vibration training in addition to a standard pulmonary rehabilitation program that includes endurance and strength training. We will include a total of 140 patients (70 patients < 1 year after lung Transplantation and 70 patients > 1 year after lung Transplantation). Our hypothesis is that an addtitional whole body vibration training produces a greater benefit to exercise capacity in lung transplantat patients (LTx).

ELIGIBILITY:
Inclusion Criteria:

* participation in an inpatient rehabilitation program
* double or single lung transplantation due to chronic obstructive pulmonary disease, Alpha-1-antitrypsine deficiency, interstitial lung disease

Exclusion Criteria:

* severe exacerbation in the last 4 weeks with the necessity of delivering antibiotics/ corticosteroids
* non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change in 6-minute walking distance | change from baseline to day 21

SECONDARY OUTCOMES:
change in Wmax | change from baseline to day 21
  maximum workload in incremental cycling test
change in Fmax | change from baseline to day 21
  maximum isometric quadriceps force
change in fibre cross sectional area | change from baseline to day 21
  cross sectional area of the M.rectus femoris, measured by ultrasound
change in chair rise time | change from baseline to day 21
  chair rise test: to get from a sitting position to a standing, measuring the time for 5 repetitions
change in quality of life | change from baseline to day 21
  SF-36 questionnaire and CRQ questionnaire
change in body cell mass | change from baseline to day 21
  measured by bio-impedance analysis
change in IGF-1 | change from baseline to day 21
  IGF-1, measured in a blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany

REFERENCES:
- [Derived] Gutierrez-Arias R, Martinez-Zapata MJ, Gaete-Mahn MC, Osorio D, Bustos L, Melo Tanner J, Hidalgo R, Seron P. Exercise training for adult lung transplant recipients. Cochrane Database Syst Rev. 2021 Jul 20;7(7):CD012307. doi: 10.1002/14651858.CD012307.pub2. PMID 34282853